CLINICAL TRIAL: NCT04188782
Title: Evaluation of the Development of Tolerance to Sevoflurane in Children Undergoing Repeated Anesthesia Exposure
Brief Title: Tolerance to Sevoflurane in Children Undergoing Repeated Drug Exposure
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Rodrigo Gutiérrez, Principal Investigator, University of Chile
Other Study IDs: 0362019
Record Dates: First submitted 2019-12-03; First posted 2019-12-06 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Anesthesia; Tolerance
Keywords: Anesthesia; Electroencephalogram; Spectral analysis
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric patients undergoing radiotherapy: Pediatric patients undergoing general anesthesia for radiotherapy treatment. General anesthesia will be accomplished exclusively by the administration of sevoflurane.
  The inhalatory induction will be performed with sevofluorane at 8% with O2 4Lt/min. The maintenance will be with sevofluorane at an end tidal of 2.5% with 1Lt/min of O2.
  The EEG will be obtain with SedLine monitor
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — Describe how a reiterative anesthesia exposure could induce tolerance to the anesthetic.

SUMMARY:
Deep sedation or general anesthesia is frequently required for infant that need radiotherapy to treat malignancies. As radiation therapy usually consist of several sessions, these patients are exposure to several consecutive anesthetic exposures (e.g. for some central nervous system tumors 30 sessions of radiotherapy are required). In our center, this 30-min anesthetic exposure are with sevoflurane. Considering that repeated daily exposure to such potent drugs, as general anesthetics, may induce tolerance, it is reasonable to explore whether this phenomenon is occurring in this population.

The aim of this observational study was to determine if a repeated exposure to sevoflurane is associated with the development of clinical and electroencephalographic tolerance.

We will enroll 16 pediatric patients, and we will measure the time needed to appropriately place the laryngeal mask (clinical effect) and we also will compare the electroencephalographic signal under anesthesia across the different sessions (electroencephalographic effect).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the development of tolerance to sevoflurane in children undergoing repeated drug exposure.

We will evaluate the development of tolerance in two ways:

Clinical: as the time needed to perform the inhalation induction, with a standardized protocol.

Electroencephalographic: we will record every 3 sessions the electroencephalographic activity of the patients. We will perform classical spectral analysis, and coherence analysis as well.

This observational study will be mainly exploratory since there are no other previous report in this topic

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radiotherapy
* Requiring general anesthesia

Exclusion Criteria:

* Previous Radiotherapy
* Malignant Hyperthermia history

Ages: 10 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All consecutive pediatric patients schedule for radiotherapy treatment under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Theta power in the EEG spectrum under anesthesia | Last session of radiotherapy (compare to first session) - Up to 6 weeks
  Theta power obtained from the EEG signal, with the patient under general anesthesia

SECONDARY OUTCOMES:
Time to Laryngeal Mask insertion | Last session of radiotherapy (compare to first session) - Up to 6 weeks
  The time in seconds between the induction beginning and the correct laryngeal mask placement
Alpha power in the EEG spectrum under anesthesia | Last session of radiotherapy (compare to first session) - Up to 6 weeks
  Alpha power obtained from the EEG signal, with the patient under general
Coherence | Last session of radiotherapy (compare to first session) - Up to 6 weeks
  Coherence between frontal electrodes in bands of the spectrum

CONTACTS AND LOCATIONS:
Overall Officials: Antonello Penna, MD PhD, Principal Investigator — University of Chile; Jose I Egaña, MD PhD, Principal Investigator — University of Chile; Felipe Maldonado, Md MSc, Principal Investigator — University of Chile; Rodrigo Gutierrez, MD PhD, Principal Investigator — University of Chile
Locations (2):
- Chile (2):
  - Instituto Nacional del Cancer, Santiago, Santiago Metropolitan
  - Centro de Investigacion Clinica Avanzada, Santiago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keidan I, Perel A, Shabtai EL, Pfeffer RM. Children undergoing repeated exposures for radiation therapy do not develop tolerance to propofol: clinical and bispectral index data. Anesthesiology. 2004 Feb;100(2):251-4. doi: 10.1097/00000542-200402000-00011. PMID 14739796